CLINICAL TRIAL: NCT04614298
Title: A Phase 4 Clinical Study to Evaluate the Efficacy and Safety of Induction and Maintenance Therapy of Brodalumab (KHK4827) in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase 4 Study of Brodalumab (KHK4827) in Subjects With Moderate to Severe Plaque Psoriasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the reconsideration of KHK4827's business in China, it. was decided to withdraw this clinical trial prior to enrollment of first participant.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4827-CN001
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK4827 210 mg SC (Subcutaneous) (Experimental): Single SC administration
  Interventions: Drug: KHK4827-Active
- Placebo SC (Placebo Comparator): Single SC administration
  Interventions: Drug: KHK4827-Placebo

INTERVENTIONS:
Drug: KHK4827-Active — Single SC administration
  Arms: KHK4827 210 mg SC (Subcutaneous)
Drug: KHK4827-Placebo — Single SC administration
  Arms: Placebo SC

SUMMARY:
The objective of this study is assessing the efficacy and safety of brodalumab in Chinese subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Those who are ≥18 and ≤70 years of age at the time of signing the written informed consent form
* Those who have involved BSA (the percentage (%) of body surface area involved with lesion) ≥10%, PASI (Psoriasis Area and Severity Index) ≥12 and sPGA (static Physician's global assessment) ≥ 3 at screening and at baseline.

Exclusion Criteria:

* Those who diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis or medication-induced psoriasis
* Those who have skin conditions other than psoriasis including eczema at the time of the screening that would interfere with evaluations of the study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of subjects achieving 75% improvement from baseline in Psoriasis Area and Severity Index (PASI; PASI 75) at Week 12 | Week 12

SECONDARY OUTCOMES:
To evaluate the proportion of subjects achieving 100% improvement from baseline in PASI (PASI 100) at Week 12 | Week 12
To evaluate static physician's global assessment (sPGA) of "clear or almost clear (0 or 1)" at Week 12 | Week 12

OTHER OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) or drug-related TEAEs | after received an investigational product until last visit 1 year

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Site 01, Beijing
  - Site 03, Beijing
  - Site 04, Beijing
  - Site 10, Beijing
  - Site 11, Beijing
  - Site 12, Beijing
  - Site 21, Beijing
  - Site 07, Changchun
  - Site 13, Changchun
  - Site 14, Chongqing
  - Site 09, Hangzhou
  - Site 17, Hangzhou
  - Site 24, Hangzhou
  - Site 25, Nanjing
  - Site 02, Shanghai
  - Site 05, Shanghai
  - Site 08, Shanghai
  - Site 06, Tianjin
  - Site 22, Tianjin
  - Site 23, Ürümqi
  - Site 16, Wenzhou
  - Site 19, Wuhan
  - Site 20, Wuhan
  - Site 15, Xi'an
  - Site 18, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided